CLINICAL TRIAL: NCT04246658
Title: Effect of Platform Swing Walkway on Locomotor Behavior in Children With Diaplegia
Brief Title: Effect of Platform Swing Walkway on Locomotor Behavior in Diplegic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hanaa mohsen (Other)
Responsible Party: Sponsor-Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hana1
Record Dates: First submitted 2020-01-15; First posted 2020-01-29 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Vestibular Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): gait training on platform swing walkway for 30 minute.
  Interventions: Other: conventional physical therapy program; Other: gait training on platform swing walkway
- control group (Experimental): conventional physical therapy program
  Interventions: Other: conventional physical therapy program

INTERVENTIONS:
Other: conventional physical therapy program — traditional physical therapy program
Other: gait training on platform swing walkway — gait training on platform swing walkway for 30 minute.
  Arms: Treatment group

SUMMARY:
Locomotor activity is accompanied by a number of sensory stimuli: visual, auditory, olfactory, vestibular, and somatosensory. When improving motor skills, incorporating postural reflexes, creating synchronized eye movements, and visual attention skills, the vestibular system is particularly important.

DETAILED DESCRIPTION:
Thirty diaplegic cerebral palsied children of both sexes, ranged in age from 3 to 6 years enrolled in this study. They randomly assigned into two groups of equal number; control group (A), study group (B). Group (A) groups received the conventional physical therapy program based on neurodevelopmental approach for such cases. Whereas study group (B) received the same conventional physical therapy program given to group (A) in addition to gait training on platform swing walkway for 30 minute. All children were assessed before and after the treatment program by using 2D video based gait assessment system to measure the percentage of swing and stance phase, also GMFM was used to assess standing and walking, running, and jumping abilities, domains (D) and (E).

ELIGIBILITY:
Inclusion Criteria:

* were cognitively competent
* able to understand and follow instructions.

Exclusion Criteria:

* if they had fixed contractures
* deformities of the spine, upper or lower extremities,
* visual or respiratory disorders.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Growth Motor Function Measure Scale (GMFM). | pre intervension and after three months of the intervention to asses the improvent in standing and walking .the highest score indicate improvementg
  Growth Motor Function Measure Scaleis the scale tat will assess the functional gross preinterventiona and after 3 months of the treatment program
2D, video based gait assessment system: | 2D, video based gait assessment system asses the change in the stance in swing phase before and after three months of the intervention program .
  Tracker Video Analysis and Modeling Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Badr Univesity in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided